CLINICAL TRIAL: NCT06285916
Title: A Randomized, Placebo-Controlled, Double-Blinded, Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of Oral NORA520 in Female Adults With Severe Postpartum Depression
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of Oral NORA520 in Adults With Severe Postpartum Depression
Acronym: NuMom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DuKang Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NORA520-PT-US-1a
Record Dates: First submitted 2024-02-17; First posted 2024-02-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Depression, Postpartum; Postpartum Depression; Post-partum Depression; Postnatal Depression; Post-Natal Depression
Keywords: Depression; Postpartum Depression; NORA520; Postnatal Depression; NuMom
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NORA520 Tablets Dose 1 (Experimental): NORA520 Tablets Dose 1
  Interventions: Drug: NORA520 Dose 1
- NORA520 Tablets Dose 2 (Experimental): NORA520 Tablets Dose 2
  Interventions: Drug: NORA520 Dose 2
- Placebo Tablets (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NORA520 Dose 1 — Oral NORA520 tablets Dose 1 for 3 days
  Arms: NORA520 Tablets Dose 1
Drug: NORA520 Dose 2 — Oral NORA520 tablets Dose 2 for 3 days
  Arms: NORA520 Tablets Dose 2
Drug: Placebo — Oral Placebo tablets for 3 days
  Arms: Placebo Tablets

SUMMARY:
The purpose of this research study is to test the study drug, NORA520, as a possible treatment for severe postpartum depression (PPD). The trial aims to determine:

* How well NORA520 is tolerated and what side effects it may cause
* If NORA520 reduces depressive symptoms in subjects with severe PPD
* The amount of NORA520 in the blood at various times after taking the study drug; this provides information that helps determine how often NORA520 should be taken
* In a subset of subjects, the amount of NORA520 in breastmilk at various times after taking it to determine if and how much NORA520 can pass into breastmilk Participate in this study will be randomly assigned to one of 3 different groups. All subjects will take the study drug for 3 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Are willing and able to provide signed informed consent to participate in the study and to comply with all study procedures and scheduled visits
* Are an adult female between 18 and 45 years of age, inclusive;
* Have either ceased lactating at Screening, or if still lactating or actively breastfeeding at Screening, agree to temporarily cease giving breastmilk to their infant(s) from just prior to first dose of study drug on Day 1 through Day 14;
* Have a negative pregnancy test at Screening and Day 1 (prior to dosing);
* Have had a depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery
* Are ≤9 months postpartum at Screening.

Key Exclusion Criteria:

* Have a history or current diagnosis or current treatment of bipolar disorder, schizophrenia, or schizoaffective disorder;
* Have had recorded treatment failure of ≥2 different antidepressant classes (e.g., SSRI, SNRI) in the current or previous episode;
* Are currently experiencing active psychosis per Investigator assessment, or are taking typical or atypical antipsychotic medication;
* Have a history of suicidal behavior within 2 years;
* Have a history or current diagnosis of sleep apnea or narcolepsy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and causality of AEs, SAEs, and AESIs | Up to Day 30
  Adverse events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs)
Change from baseline in HAM-D17 total score compared to placebo | Baseline to Day 4
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) contains 17 individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia (initial, middle, and late), work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic and somatic), gastrointestinal symptoms, general somatic symptoms, sexual interest, hypochondriasis, insight, and weight loss. The total score ranges from 0 to 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change from baseline in HAM-D17 total score | Baseline to Days 8 and 30
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) contains 17 individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia (initial, middle, and late), work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic and somatic), gastrointestinal symptoms, general somatic symptoms, sexual interest, hypochondriasis, insight, and weight loss. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17 response | Baseline to Days 4, 8, and 30
  Defined as having a 50% or greater reduction from baseline in HAM-D17 total score. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17 remission | Baseline to Days 4, 8, and 30
  Defined as having a HAM-D17 total score ≤7. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
Change from baseline in HAM-D17 subscale and individual item scores | Baseline to Days 4, 8, and 30
  The Seventeen-Item Hamilton Rating Scale for Depression (HAM-D17) contains 17 individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia (initial, middle, and late), work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic and somatic), gastrointestinal symptoms, general somatic symptoms, sexual interest, hypochondriasis, insight, and weight loss. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
Change from baseline in Clinical Global Impression - Severity (CGI-S) score | Baseline to Days 4, 8, and 30
  The CGI-S scale is a 7-point scale that requires the Investigator to assess how mentally ill is the patient at this time. 1 - normal, not at all ill; 2 - borderline mentally ill; 3 - mildly ill; 4 - moderately ill; 5 - markedly ill; 6 - severely ill; or 7 - among the most extremely ill patients.
Clinical Global Impression - Improvement (CGI-I) scale positive response | Baseline to Days 4, 8, and 30
  The CGI-I scale is a 7-point scale that requires the Investigator to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of study drug treatment. 1 - very much improved; 2 - much improved; 3 - minimally improved; 4 - no change; 5 - minimally worse; 6 - much worse; or 7 - very much worse
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) total score | Baseline to Days 4, 8, and 30
  The MADRS contains 10 individual items related to the following symptoms: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The total score ranges from 0 to 60, with higher scores indicating more severe depression.
Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) total score | Baseline to Days 4, 8, and 30
  The HAM-A contains 14 individual ratings related to the following symptoms: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic (muscular), somatic (sensory), cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. The total score ranges from 0 to 56, with higher scores indicating more severe anxiety.
Change from baseline in Edinburgh Postnatal Depression Scale (EPDS) total score | Baseline to Days 8 and 30
  The Edinburgh Postnatal Depression Scale (EPDS) is a set of 10 screening questions. The total score ranges from 0 to 30, with higher scores indicating more severe depression.
Number of patients who start any new antidepressant or anti-anxiety medication | After Day 8 assessments through Day 30

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Advanced Research Center, Anaheim, California
  - Alliance Research Institute, Canoga Park, California
  - Cenexel Clinical Research, Sherman Oaks, California
  - Cenexel Clinical Research, Torrance, California
  - MedOne Clinical Research, Miami, Florida
  - Meridian International Research, Inc., Miami Gardens, Florida
  - Combined Research, Orlando, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - GCP Research, St. Petersburg, Florida
  - Cenexel Clinical Research, Atlanta, Georgia
  - CenExel Clinical Research, Decatur, Georgia
  - CenExel Clinical Research, Savannah, Georgia
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - Zucker Hillside Hospital, Glen Oaks, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Maximos Ob/Gyn, League City, Texas
  - Pillar Clinical Researc, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No